CLINICAL TRIAL: NCT00828841
Title: A Multi-Center Randomized Phase 2b Study of Cetuximab (Erbitux) in Combination With Platinum-Based Chemotherapy as First Line Treatment of Patients With Recurrent or Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase 2b Study of Cetuximab With Platinum-Based Chemo as First Line Treatment of Recurrent or Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC01L08
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Paclitaxel; Carboplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paclitaxel, Carboplatin, Cetuximab (Arm A) (Active Comparator): Patients with squamous or non-squamous histologies will receive carboplatin and paclitaxel for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion.
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Carboplatin
- Platinum, Gemcitabine, Cetuximab (Arm B) (Active Comparator): Patients with squamous or non-squamous histologies will receive gemcitabine with either carboplatin or cisplatin for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion. The choice of platinum-based chemotherapy is also at the investigator's discretion.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: Gemcitabine; Drug: Cisplatin
- Platinum, Pemetrexed, Cetuximab (Arm C) (Active Comparator): Patients with squamous histology will receive pemetrexed and either carboplatin or cisplatin for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion. The choice of platinum-based chemotherapy is also at the investigator's discretion. Patients with non-squamous histology are not eligible for this arm.
  Interventions: Drug: Cetuximab; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be administered at a loading dose of 400 mg/m2 on Day 1, Cycle 1 and at a dose of 250 mg/m2 weekly during chemotherapy. During the maintenance period, cetuximab will be dosed at 500 mg/m2 every two weeks.
  Other Names: Erbitux
Drug: Paclitaxel — Paclitaxel 200 mg/m2 Day 1 every 21 days
  Other Names: Taxol
  Arms: Paclitaxel, Carboplatin, Cetuximab (Arm A)
Drug: Carboplatin — Carboplatin AUC 6 Day 1 every 21 days
  Other Names: Paraplatin
Drug: Gemcitabine — Gemcitabine 1,000 mg/m2 Days 1 and 8 every 21 days
  Other Names: Gemzar
  Arms: Platinum, Gemcitabine, Cetuximab (Arm B)
Drug: Cisplatin — Cisplatin 75 mg/m2 Day I every 21 days
  Other Names: Platinol
  Arms: Platinum, Gemcitabine, Cetuximab (Arm B); Platinum, Pemetrexed, Cetuximab (Arm C)

SUMMARY:
This study is testing the investigational drug, cetuximab, in combination with different chemotherapy drugs for lung cancer. The aim of the study is to determine which of the drug combinations looks most promising and should be tested further. The study will also look at what side effects may occur.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before study-related activities
* Histologically or cytologically confirmed Stage IIIb with cytologically documented malignant pleural or pericardial effusion, Stage IV, or recurrent non-smal cell lung cancer (NSCLC) after resection or radiation for earlier stage disease
* Measurable or evaluable disease (per modified Response Evaluation Criteria in Solid Tumors [RECIST] guidelines)
* Male or female ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* White blood count ≥ 3 x 10(9)/L with neutrophils ≥ 1.5 x 10(9)/L, platelet count ≥ 100 x 10(9)/L, and hemoglobin ≥ 9.5 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5 x ULN in patients with liver mets
* Serum creatinine ≤ 1.25 x ULN
* Recovery from prior surgery or radiation to Grade 1 or better toxicity
* Women of childbearing potential (WOCBP) and fertile men with partners of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 wks after the study in such a manner that the risk of pregnancy is minimized
* WOCBP must have a negative serum or urine pregnancy test within 72 hrs prior to the start of study medication or in accordance with local regulations, whichever is of shorter duration

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test during screening or prior to study drug administration
* Sexually active fertile men not using effective birth control if their partners are women of child-bearing potential
* Prior chemo for advanced NSCLC; neoadjuvant or post-operative adjuvant chemo is allowed if completed at least 12 months before study entry
* Previous exposure to epidermal growth factor receptor (EGFR)-targeted therapy. Prior treatment with monoclonal antibodies targeting receptors other than the EGFR, such as bevacizumab, is allowed if completed > 30 days prior to randomization
* Treatment with any investigational agent(s) within 4 weeks prior to study entry
* Concurrent anti-cancer therapy (chemotherapy, hormonal therapy, biologic or targeted therapy) other than protocol therapy
* Carcinoid, atypical carcinoid or small cell lung cancer
* Symptomatic or uncontrolled mets in the central nervous system
* Prior invasive malignancy requiring ongoing therapy within the past year
* Active infection (infection requiring intravenous [IV] antibiotics), including active tuberculosis, known and declared HIV
* Myocardial infarction within 6 months prior to study entry, uncontrolled congestive heart failure; or any current Grade 3 or 4 cardiovascular disorder despite treatment
* Known allergic/hypersensitivity reaction to any of the components of study treatments
* Peripheral neuropathy ≥ Grade 2, as assessed by Common Terminology Criteria for Adverse Events, version 3.0
* History of significant neurologic or psychiatric disorders including but not limited to dementia, seizures, and bipolar disorder
* Medical or psychological condition that would not permit the patient to complete the study or sign informed consent
* Known drug abuse

Patients of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Schwartzberg, MD, FACP, Study Chair — Accelerated Community Oncology Research Network
Locations (84):
- United States (84):
  - Anniston, Alabama
  - Jonesboro, Arkansas
  - Anaheim, California
  - Azusa, California
  - Burbank, California
  - Campbell, California
  - Greenbrae, California
  - Hawthorne, California
  - Mission Hills, California
  - Orange, California
  - Oxnard, California
  - St. Helena, California
  - Fort Collins, Colorado
  - Norwich, Connecticut
  - Torrington, Connecticut
  - Trumbull, Connecticut
  - Fort Lauderdale, Florida
  - Lake Worth, Florida
  - Orange City, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Titusville, Florida
  - Weston, Florida
  - Augusta, Georgia
  - Columbus, Georgia
  - Lawrenceville, Georgia
  - Marietta, Georgia
  - Valdosta, Georgia
  - Elmhurst, Illinois
  - Harvey, Illinois
  - Joliet, Illinois
  - Quincy, Illinois
  - Skokie, Illinois
  - South Bend, Indiana
  - Family Medicine of Vincennes, Vincennes, Indiana
  - Arnes, Iowa
  - Bettendorf, Iowa
  - Mason City, Iowa
  - Waterloo, Iowa
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Lafayette, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Towson, Maryland
  - Springfield, Massachusetts
  - Worchester, Massachusetts
  - Jefferson City, Missouri
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Portsmouth, New Hampshire
  - Bellville, New Jersey
  - Cherry Hill, New Jersey
  - Elizabeth, New Jersey
  - Hackensack, New Jersey
  - East Setauket, New York
  - Fresh Meadows, New York
  - The Bronx, New York
  - Fayetteville, North Carolina
  - Gastonia, North Carolina
  - Goldsboro, North Carolina
  - Columbus, Ohio
  - Dayton, Ohio
  - Middletown, Ohio
  - Sandusky, Ohio
  - Bend, Oregon
  - Bethlehem, Pennsylvania
  - Reading, Pennsylvania
  - Sumter, South Carolina
  - Sioux Falls, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Lubbock, Texas
  - Bennington, Vermont
  - Kirkland, Washington
  - Tacoma, Washington
  - Huntington, West Virginia
  - Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to enrollment at 118 oncology clinics from November 2008 to May 2011.
Pre-assignment Details: Consent was obtained from all subjects. Subjects were stratified by histology (non-squamous vs. squamous), followed by disease stage (IIIb vs. IV). Subjects in the non-squamous stratum were randomized to 1 of 3 treatment arms (Arm A, B, or C); subjects in the squamous stratum were randomized to only 1 of 2 of these treatment arms (Arm A or B).
Groups:
- Paclitaxel, Carboplatin, Cetuximab (Arm A): Patients with squamous or non-squamous histologies will receive carboplatin and paclitaxel for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion.
  Paclitaxel : Paclitaxel 200 mg/m2 Day 1 every 21 days
  Carboplatin : Carboplatin AUC 6 Day 1 every 21 days
  Cetuximab : Cetuximab will be administered at a loading dose of 400 mg/m2 on Day 1, Cycle 1 and at a dose of 250 mg/m2 weekly during chemotherapy. During the maintenance period, cetuximab will be dosed at 500 mg/m2 every two weeks.
- Platinum, Gemcitabine, Cetuximab (Arm B): Patients with squamous or non-squamous histologies will receive gemcitabine with either carboplatin or cisplatin for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion. The choice of platinum-based chemotherapy is also at the investigator's discretion.
  Gemcitabine : Gemcitabine 1,000 mg/m2 Days 1 and 8 every 21 days
  Cisplatin : Cisplatin 75 mg/m2 Day I every 21 days
  Carboplatin : Carboplatin AUC 6 Day 1 every 21 days
  Cetuximab : Cetuximab will be administered at a loading dose of 400 mg/m2 on Day 1, Cycle 1 and at a dose of 250 mg/m2 weekly during chemotherapy. During the maintenance period, cetuximab will be dosed at 500 mg/m2 every two weeks.
- Platinum, Pemetrexed, Cetuximab (Arm C): Patients with squamous histology will receive pemetrexed and either carboplatin or cisplatin for a minimum of four and a maximum of six 21-day cycles, plus cetuximab, and then enter a maintenance phase with single-agent cetuximab. Cetuximab will be given on Day 1, and weekly during chemotherapy, followed by biweekly administration during the maintenance period. The choice of delivering four, five or six cycles of chemotherapy is at the investigator's discretion. The choice of platinum-based chemotherapy is also at the investigator's discretion. Patients with non-squamous histology are not eligible for this arm.
  Cisplatin : Cisplatin 75 mg/m2 Day I every 21 days
  Carboplatin : Carboplatin AUC 6 Day 1 every 21 days
  Cetuximab : Cetuximab will be administered at a loading dose of 400 mg/m2 on Day 1, Cycle 1 and at a dose of 250 mg/m2 weekly during chemotherapy. During the maintenance period, cetuximab will be dosed at 500 mg/m2 every two weeks.
Period: Overall Study
Arm/Group | Paclitaxel, Carboplatin, Cetuximab (Arm A) | Platinum, Gemcitabine, Cetuximab (Arm B) | Platinum, Pemetrexed, Cetuximab (Arm C)
Started | 235 | 236 | 130
Completed | 231 | 232 | 126
Not Completed | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel, Carboplatin, Cetuximab (Arm A) | Platinum, Gemcitabine, Cetuximab (Arm B) | Platinum, Pemetrexed, Cetuximab (Arm C) | Total
Number analyzed (Participants) | 235 | 236 | 130 | 601
Age Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.9) | 64.9 (9.5) | 65.6 (9.4) | 65.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 90 | 64 | 251
  Male | 138 | 146 | 66 | 350
Region of Enrollment [Number; unit: participants]
  United States | 235 | 236 | 130 | 601

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival by Treatment Arm
Time Frame: Survival was measured from the date of randomization to date of death due to any cause, assessed up to 36 months. Subjects who were alive at the date of last contact were censored at the date of last contact.
Population: Two subjects in Arm A were censored due to negative event intervals.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel, Carboplatin, Cetuximab (Arm A) | Platinum, Gemcitabine, Cetuximab (Arm B) | Platinum, Pemetrexed, Cetuximab (Arm C)
Number analyzed (Participants) | 233 | 236 | 130
Months | 9.5 [8.3 to 11.4] | 8.3 [7.1 to 9.9] | 10.6 [8.0 to 14.5]

2. Secondary Outcome: 1-year Survival by Treatment Arm
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel, Carboplatin, Cetuximab (Arm A) | Platinum, Gemcitabine, Cetuximab (Arm B) | Platinum, Pemetrexed, Cetuximab (Arm C)
Number analyzed (Participants) | 233 | 236 | 130
percentage of participants | 39.7 [33.7 to 46.6] | 37.2 [31.3 to 44.2] | 47.3 [39.1 to 57.1]

3. Secondary Outcome: Overall Survival by Histology
Time Frame: as for outcome 1
Population: Subjects were stratified by histology prior to randomization to a treatment arm.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Squamous Cell Histology: Subjects who were identified as having squamous cell histology, prior to randomization to a treatment arm.
- Non-squamous Cell Histology: Subjects who were identified as having non-squamous cell histology, prior to randomization to a treatment arm.
Arm/Group | Squamous Cell Histology | Non-squamous Cell Histology
Number analyzed (Participants) | 200 | 399
Months | 8.7 [7.4 to 10.1] | 9.9 [8.3 to 11.4]

ADVERSE EVENTS:
Time Frame: Adverse events collection began at the time the patient signed the informed consent and continued throughout the study until 30 days after the last dose.
Description: Systematic Assessment - subjects were assessed for adverse events by a member of the research team every 1-2 weeks.
Arm/Group | Paclitaxel, Carboplatin, Cetuximab (Arm A) | Platinum, Gemcitabine, Cetuximab (Arm B) | Platinum, Pemetrexed, Cetuximab (Arm C)
Serious Adverse Events (participants affected / at risk) | 109/235 | 128/236 | 68/130
Other Adverse Events (participants affected / at risk) | 221/235 | 215/236 | 119/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Carboplatin, Cetuximab (Arm A) (N=235) | Platinum, Gemcitabine, Cetuximab (Arm B) (N=236) | Platinum, Pemetrexed, Cetuximab (Arm C) (N=130)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Accidental Exposure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 3 | 0
Adverse Reation (General disorders) | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 2 | 6 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 19 | 6
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arterial Thrombosis (Vascular disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 4 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Bacteremia (Infections and infestations) | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Blood/Bone Marrow Hemoglobin (Investigations) | 0 | 0 | 1
Brain Edema (Nervous system disorders) | 0 | 1 | 0
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 2 | 1
Catheter Site Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 2
Central Nervous System Hemorrhage (Nervous system disorders) | 1 | 0 | 1
Central Pain Syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 3 | 3 | 1
Chest Pain (General disorders) | 6 | 5 | 1
Chills (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Clostridial Infection (Infections and infestations) | 2 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Convulsion (Nervous system disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cytokine Release Syndrome (Immune system disorders) | 0 | 1 | 0
Death (General disorders) | 5 | 3 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Deep Vein Thrombosis (Vascular disorders) | 4 | 9 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 8 | 7
Depression (Psychiatric disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 1
Disease Progression (General disorders) | 5 | 7 | 6
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 6
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Eastern Cooperative Oncology Group Performance Status (Investigations) | 0 | 1 | 1
Ejection Fraction Decreased (Investigations) | 0 | 1 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 0 | 1
Esophageal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 2
Fungemia (Infections and infestations) | 0 | 0 | 1
Gastric Ulcer Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 | 3 | 2
General Physical Health Deterioration (General disorders) | 0 | 1 | 0
Generalized Edema (General disorders) | 1 | 0 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hemoglobin (Investigations) | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 4 | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 5 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1
Infection (Infections and infestations) | 3 | 0 | 0
Infectious Pleural Effusion (Infections and infestations) | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 8 | 2 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Large Cell Carcinoma Of The Respiratory Tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Leg Amputation (Surgical and medical procedures) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lipase Increased (Investigations) | 1 | 0 | 0
Lung Infection (Immune system disorders) | 0 | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Medication Error (Injury, poisoning and procedural complications) | 0 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 3 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 3 | 0
Myocardial Ischemia (Cardiac disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0 | 0
Neutrophil Count (Investigations) | 1 | 1 | 2
Neutrophil Count Decreased (Investigations) | 1 | 1 | 0
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 3 | 2
Pericardial Effusion Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peripheral Edema (General disorders) | 1 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 5
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 15 | 9 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 3
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 1
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 1 | 1 | 0
Recall Phenomenon (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 2 | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Restrictive Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 0 | 4
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0
Spinal Pain (General disorders) | 1 | 0 | 0
Splenic Hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 1
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subdural Hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Superior Vena Cava Syndrome (Vascular disorders) | 1 | 0 | 2
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 3 | 3
Tachycardia (Cardiac disorders) | 3 | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 15 | 3
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0
Transient Ischemic Attack (Nervous system disorders) | 1 | 0 | 0
Troponin Increased (Investigations) | 0 | 0 | 1
Tumor Embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ulcer Hemorrhage (General disorders) | 1 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Urinart Tract Infection (Infections and infestations) | 2 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
Venous Valve Ruptured (Vascular disorders) | 0 | 1 | 0
Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3
White Blood Cell Count (Investigations) | 1 | 0 | 0
White Blood Cell Increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Carboplatin, Cetuximab (Arm A) (N=235) | Platinum, Gemcitabine, Cetuximab (Arm B) (N=236) | Platinum, Pemetrexed, Cetuximab (Arm C) (N=130)
7th Nerve Paralysis (Nervous system disorders) | 1 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 19 | 18 | 7
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 5 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 6 | 4
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 1
Abscess Drainage (Surgical and medical procedures) | 0 | 1 | 0
Abscess Neck (Infections and infestations) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 1
Adrenal Mass (Endocrine disorders) | 0 | 1 | 0
Adverse Drug Reaction (General disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 3 | 2
Alanine Aminotransferase (Investigations) | 1 | 3 | 3
Alanine Aminotransferase Decreased (Investigations) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 10 | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 27 | 6
Amylase Increased (Investigations) | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 83 | 105 | 52
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Anhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 17 | 17 | 9
Aortic Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 15 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate Aminotransferase (Investigations) | 2 | 2 | 2
Aspartate Aminotransferase Increased (Investigations) | 8 | 10 | 7
Asthenia (General disorders) | 24 | 13 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 4 | 0
Atrial Septal Defect Repair (Surgical and medical procedures) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 25 | 21
Bacterial Sepsis (Infections and infestations) | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 1 | 2 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Biopsy Endometrium (Investigations) | 0 | 1 | 0
Bladder Pain (Renal and urinary disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 2 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0
Blindness (Eye disorders) | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood Albumin (Investigations) | 0 | 1 | 1
Blood Albumin Decreased (Investigations) | 5 | 4 | 1
Blood Alkaline Phosphatase (Investigations) | 7 | 6 | 4
Blood Alkaline Phosphatase Decreased (Investigations) | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 18 | 14 | 6
Blood Bicarbonate Abnormal (Investigations) | 0 | 0 | 1
Blood Bicarbonate Decreased (Investigations) | 2 | 0 | 1
Blood Bilirubin Decreased (Investigations) | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 2 | 1
Blood Calcium Decreased (Investigations) | 2 | 3 | 1
Blood Chloride Decreased (Investigations) | 2 | 1 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 2
Blood Creatinine (Investigations) | 0 | 1 | 3
Blood Creatinine Decreased (Investigations) | 1 | 1 | 0
Blood Creatinine Increased (Investigations) | 3 | 4 | 3
Blood Electrolytes Decreased (Investigations) | 1 | 0 | 0
Blood Glucose (Investigations) | 1 | 1 | 1
Blood Glucose Decreased (Investigations) | 2 | 1 | 0
Blood Glucose Increased (Investigations) | 5 | 4 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 1
Blood Magnesium (Investigations) | 0 | 2 | 1
Blood Magnesium Decreased (Investigations) | 18 | 10 | 9
Blood Phosphorus Decreased (Investigations) | 1 | 0 | 1
Blood Potassium (Investigations) | 1 | 1 | 1
Blood Potassium Decreased (Investigations) | 0 | 5 | 1
Blood Potassium Increased (Investigations) | 1 | 0 | 1
Blood Pressure Decreased (Investigations) | 1 | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 0 | 0
Blood Sodium (Investigations) | 1 | 0 | 0
Blood Sodium Decreased (Investigations) | 1 | 2 | 1
Blood Sodium Increased (Investigations) | 3 | 0 | 0
Blood Urea Decreased (Investigations) | 5 | 2 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 1
Blood Uric Acid Increased (Investigations) | 1 | 0 | 0
Blood/Bone Marrow Hemoglobin (Investigations) | 0 | 1 | 2
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 17 | 7 | 3
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Breath Sounds Abnormal (Investigations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 5 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Burning Sensation (Nervous system disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Candidiasis (Infections and infestations) | 3 | 3 | 6
Carbuncle (Infections and infestations) | 1 | 0 | 0
Cardiac Valve Disease (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Catheter Placement (Surgical and medical procedures) | 1 | 2 | 0
Catheter Site Discharge (General disorders) | 0 | 1 | 0
Catheter Site Erythema (General disorders) | 0 | 2 | 1
Catheter Site Infection (Infections and infestations) | 0 | 1 | 0
Catheter Site Pain (General disorders) | 2 | 3 | 1
Cellulitis (Infections and infestations) | 2 | 3 | 3
Central Nervous System Hemorrhage (Nervous system disorders) | 0 | 1 | 0
Central Venous Catheterization (Surgical and medical procedures) | 0 | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 1
Chemical Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest Discomfort (General disorders) | 3 | 3 | 1
Chest Pain (General disorders) | 13 | 18 | 10
Chest Wall Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chest X-Ray Abnormal (Investigations) | 0 | 0 | 1
Chills (General disorders) | 9 | 14 | 4
Cholelithotomy (Surgical and medical procedures) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Coagulation Factor Decreased (Investigations) | 1 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 1 | 0
Colony Stimulating Factor Therapy (Surgical and medical procedures) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 14 | 7 | 4
Conjunctival Hemorrhage (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 4 | 3 | 5
Conjunctivitis Infective (Infections and infestations) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 79 | 75 | 39
Contusion (Injury, poisoning and procedural complications) | 6 | 4 | 4
Convulsion (Nervous system disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 52 | 22
Cushingoid (Endocrine disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Dark Circles Under Eyes (Eye disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 3 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 74 | 63 | 44
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 5 | 4 | 1
Deep Vein Thrombosis (Vascular disorders) | 7 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 29 | 19 | 12
Depression (Psychiatric disorders) | 17 | 11 | 9
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 1 | 4
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 68 | 55 | 32
Device Infusion Issue (General disorders) | 0 | 0 | 1
Device Malfunction (General disorders) | 1 | 0 | 0
Device Occlusion (General disorders) | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 70 | 47 | 25
Diplopia (Eye disorders) | 1 | 3 | 0
Disease Progression (General disorders) | 1 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 26 | 32 | 22
Drug Hypersensitivity (Immune system disorders) | 6 | 3 | 1
Drug Hypersensitivity (General disorders) | 0 | 1 | 0
Dry Eye (Eye disorders) | 2 | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 4 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 27 | 31 | 13
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 21 | 24 | 3
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 11 | 8
Dysphagia (Gastrointestinal disorders) | 7 | 8 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 62 | 74 | 36
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 13 | 6
Dysuria (Renal and urinary disorders) | 3 | 7 | 2
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Ear Disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 2
Ear Pain (Ear and labyrinth disorders) | 1 | 1 | 0
Early Satiety (General disorders) | 0 | 1 | 0
Eastern Cooperative Oncology Group Performance Status (Investigations) | 44 | 39 | 31
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Edema (General disorders) | 4 | 2 | 4
Effusion (General disorders) | 1 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 | 33 | 16
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 5
Esophageal Candidiasis (Infections and infestations) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 2 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 4
Extravasation (General disorders) | 0 | 0 | 1
Eye Infection (Infections and infestations) | 0 | 0 | 2
Eye Inflammation (Eye disorders) | 0 | 1 | 0
Eye Irritation (Eye disorders) | 1 | 2 | 2
Eye Pruritus (Eye disorders) | 0 | 0 | 2
Eye Ptosis (Eye disorders) | 1 | 1 | 0
Eye Swelling (Eye disorders) | 0 | 1 | 0
Face Edema (General disorders) | 0 | 1 | 0
Facial Paresis (Nervous system disorders) | 0 | 0 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0
Fatigue (General disorders) | 131 | 131 | 76
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Feces Discolored (Gastrointestinal disorders) | 0 | 2 | 1
Feces Hard (Gastrointestinal disorders) | 1 | 0 | 0
Feeling Hot (General disorders) | 0 | 2 | 0
Feeling Jittery (General disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 5 | 4
Flushing (Vascular disorders) | 4 | 7 | 2
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 2 | 2 | 1
Furuncle (Infections and infestations) | 2 | 0 | 2
Gait Disturbance (General disorders) | 1 | 1 | 0
Gamma-Glutamyltransferase (Investigations) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis Hemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 6 | 5 | 3
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 0
General Symptom (General disorders) | 0 | 1 | 0
Genital Burning Sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Hair Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Hallucination (Psychiatric disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 26 | 25 | 19
Heart Rate Irregular (Investigations) | 1 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Hematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Hematocrit (Investigations) | 0 | 0 | 1
Hematocrit Decreased (Investigations) | 0 | 1 | 1
Hematology Test Abnormal (Investigations) | 0 | 1 | 0
Hematoma (Vascular disorders) | 3 | 0 | 0
Hematuria (Renal and urinary disorders) | 3 | 3 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 2
Hemoglobin (Investigations) | 16 | 17 | 12
Hemoglobin Decreased (Investigations) | 11 | 21 | 7
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 4
Hemorrhage (Vascular disorders) | 0 | 1 | 0
Hemorrhage Diathesis (Blood and lymphatic system disorders) | 1 | 0 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 4 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 8 | 4
Hepatic Enzyme Increased (Investigations) | 0 | 2 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hernia (General disorders) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 2 | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 1 | 1 | 3
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperbiliubinemia (Hepatobiliary disorders) | 2 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 7 | 3
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23 | 15 | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 5 | 4
Hyperlipidemia (Investigations) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 5
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hyperreflexia (Nervous system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 10 | 4 | 2
Hypersensitivity (General disorders) | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 3 | 7
Hypertriglyceridemia (Investigations) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 2 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 18 | 9
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 16 | 13
Hypoesthesia (Nervous system disorders) | 8 | 4 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 4 | 3
Hypokalemia (Metabolism and nutrition disorders) | 34 | 24 | 22
Hypomagnesemia (Metabolism and nutrition disorders) | 80 | 64 | 37
Hyponatremia (Metabolism and nutrition disorders) | 17 | 18 | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypotension (Vascular disorders) | 29 | 14 | 10
Hypothermia (General disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Hypovolemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 3
Implant Site Scar (General disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 3 | 1
Inflammatory Pain (General disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 1 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 12 | 13 | 4
Infusion Site Extravasation (General disorders) | 0 | 1 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Injection Site Reaction (General disorders) | 1 | 0 | 0
Inner Ear Disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 31 | 32 | 16
Intermittent Claudication (Vascular disorders) | 1 | 0 | 0
International Normalized Ratio Decreased (Investigations) | 0 | 1 | 1
International Normalized Ratio Increased (Investigations) | 3 | 3 | 0
Intervertebral Disc Protusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intestinal Mass (Gastrointestinal disorders) | 1 | 1 | 0
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Ischemia (Vascular disorders) | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Kawasaki's Disease (Vascular disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 2 | 2
Lacrimation Increased (Eye disorders) | 3 | 8 | 8
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 1 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 20 | 20 | 13
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lip Dry (Gastrointestinal disorders) | 1 | 0 | 0
Lip Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lip Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Local Swelling (General disorders) | 1 | 0 | 0
Localized Edema (General disorders) | 1 | 3 | 1
Localized Infection (Infections and infestations) | 4 | 6 | 1
Loss Of Consciousness (Nervous system disorders) | 2 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 2 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lyme Disease (Infections and infestations) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphatic Disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0 | 0
Lymphocyte Count (Investigations) | 4 | 3 | 1
Lymphocyte Count Decreased (Investigations) | 2 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 19 | 18 | 20
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Magnesium Metabolism Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 2 | 1 | 0
Mass (General disorders) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Medical Device Change (Surgical and medical procedures) | 0 | 1 | 0
Memory Impairment (Nervous system disorders) | 5 | 2 | 3
Mental Status Changes (Psychiatric disorders) | 3 | 0 | 0
Metabolic Function Test (Investigations) | 1 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 1 | 0
Middle Ear Effusion (Ear and labyrinth disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 2 | 0
Mouth Hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Mucosal Inflammation (General disorders) | 25 | 12 | 21
Muscle Contractions Involuntary (Nervous system disorders) | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 9 | 12 | 13
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 9 | 11 | 9
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 15 | 9 | 3
Myalgia (General disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 5 | 3
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nail Bed Infection (Infections and infestations) | 0 | 0 | 1
Nail Bed Inflammation (Infections and infestations) | 0 | 1 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 8 | 5 | 2
Nail Infection (Infections and infestations) | 1 | 0 | 0
Nail Operation (Surgical and medical procedures) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Nasal Discharge Discoloration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 98 | 84 | 61
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4
Nervousness (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 2 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 54 | 11 | 4
Neutropenia (Blood and lymphatic system disorders) | 79 | 91 | 42
Neutrophil Count (Investigations) | 14 | 17 | 10
Neutrophil Count Decreased (Investigations) | 12 | 11 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Nocturia (Renal and urinary disorders) | 0 | 2 | 0
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0
Occult Blood Positive (Investigations) | 0 | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Optic Nerve Sheath Hemorrhage (Eye disorders) | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 4 | 5 | 3
Oral Discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 0 | 2
Oral Infection (Infections and infestations) | 0 | 0 | 1
Oral Mucosal Erythema (Gastrointestinal disorders) | 1 | 0 | 1
Oral Pain (Gastrointestinal disorders) | 3 | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 3
Orthostatic Hypotension (Vascular disorders) | 3 | 1 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 1 | 0
Otitis Media (Infections and infestations) | 2 | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1
Pain (General disorders) | 23 | 16 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 25 | 16 | 10
Pain Of Skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 | 3 | 3
Palpitations (Cardiac disorders) | 2 | 2 | 4
Pancytopenia (Blood and lymphatic system disorders) | 2 | 10 | 3
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 7 | 2 | 8
Paresthesia Oral (Gastrointestinal disorders) | 1 | 0 | 0
Paronychia (Infections and infestations) | 11 | 3 | 7
Parotitis (Infections and infestations) | 0 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Penile Swelling (Reproductive system and breast disorders) | 0 | 0 | 1
Penile Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Performance Status Decreased (General disorders) | 0 | 0 | 1
Perianal Erythema (Gastrointestinal disorders) | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 1 | 0
Perineal Abscess (Infections and infestations) | 1 | 1 | 0
Periorbital Edema (Eye disorders) | 1 | 0 | 0
Peripheral Edema (General disorders) | 26 | 34 | 12
Peripheral Embolism (Vascular disorders) | 0 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 1 | 2
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 36 | 6 | 4
Peroneal Nerve Palsy (Nervous system disorders) | 2 | 0 | 0
Personality Change (Psychiatric disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 8 | 1
Phantom Pain (Nervous system disorders) | 1 | 0 | 0
Pharyngitis Bacterial (Infections and infestations) | 1 | 0 | 0
Phlebitis Superficial (Vascular disorders) | 0 | 1 | 1
Photopsia (Eye disorders) | 0 | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Platelet Count (Investigations) | 7 | 15 | 8
Platelet Count Decreased (Investigations) | 7 | 22 | 7
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pleurodesis (Surgical and medical procedures) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 9 | 3 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 3
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 3
Protein Total Decreased (Investigations) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 22 | 2
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 23 | 23 | 10
Radiation Mucositis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 88 | 100 | 51
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Raynaud's Phenomenon (Vascular disorders) | 0 | 1 | 0
Recall Phenomenon (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 4 | 2
Red Blood Cell Count Decreased (Investigations) | 0 | 1 | 0
Reflux Gastritis (Gastrointestinal disorders) | 1 | 2 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 2 | 3 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 5
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Saliva Altered (Gastrointestinal disorders) | 1 | 0 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scrotal Infection (Infections and infestations) | 0 | 0 | 1
Sensation of Pressure (General disorders) | 0 | 1 | 0
Sensory Loss (Nervous system disorders) | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Sinus Headache (Nervous system disorders) | 0 | 2 | 0
Sinus Operation (Surgical and medical procedures) | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 3 | 3 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 0
Skin Atrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Candida (Infections and infestations) | 0 | 0 | 1
Skin Depigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Skin Infection (Infections and infestations) | 0 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin Lesion Excision (Surgical and medical procedures) | 0 | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1
Slow Speech (Nervous system disorders) | 0 | 1 | 0
Soft Tissue Inflammation (General disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 1
Sputum Discolored (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Staphylococcal Bacteremia (Infections and infestations) | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Staphylococcus Test Positive (Investigations) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 24 | 20 | 14
Stool Ph Decreased (Investigations) | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Subcutaneous Abscess (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subdural Hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 2
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 5 | 4 | 2
Tachycardia (Cardiac disorders) | 9 | 11 | 3
Tearfulness (Psychiatric disorders) | 0 | 0 | 1
Temperature Intolerance (General disorders) | 1 | 1 | 0
Tenderness (General disorders) | 2 | 2 | 0
Tension Headache (Nervous system disorders) | 0 | 1 | 0
Therapy Regimen Changed (Surgical and medical procedures) | 1 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 61 | 122 | 49
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2 | 1
Tinea Cruris (Infections and infestations) | 0 | 1 | 0
Tinea Pedis (Infections and infestations) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 4 | 6 | 2
Tongue Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 11 | 4
Trichomegaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1 | 0
Troponin I Increased (Investigations) | 0 | 1 | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Upper Aerodigestive Tract Infection (Infections and infestations) | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 6 | 4
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Urinary Bladder Hemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 9 | 9 | 7
Urine Color Abnormal (Investigations) | 0 | 1 | 0
Urine Flow Decreased (Renal and urinary disorders) | 0 | 1 | 0
Urine Output Decreased (Investigations) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 2
Vaginal Infection (Infections and infestations) | 1 | 0 | 0
Venous Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Venous Insufficiency (Vascular disorders) | 0 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0
Vision Blurred (Eye disorders) | 7 | 7 | 3
Visual Impairment (Eye disorders) | 3 | 2 | 3
Vitamin B12 Deficiency (Investigations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 41 | 47 | 27
Vulvitis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal Erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 2 | 2 | 0
Weight (Investigations) | 1 | 1 | 1
Weight Decreased (Investigations) | 119 | 100 | 56
Weight Fluctuation (Metabolism and nutrition disorders) | 3 | 5 | 2
Weight Increased (Investigations) | 26 | 23 | 13
Weight Normal (Investigations) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3
White Blood Cell Count (Investigations) | 14 | 16 | 16
White Blood Cell Count Decreased (Investigations) | 2 | 6 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 1
White Blood Cell Disorder (Blood and lymphatic system disorders) | 3 | 4 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Xerophthalmia (Eye disorders) | 0 | 0 | 1
Xerosis (General disorders) | 0 | 0 | 1
Tobacco User (Social circumstances) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study funder will be provided with a copy of any results communication at least 30 days prior to its submission to a scientific journal or presentation at a scientific meeting to allow review of the publication for confidential information. If confidential information is being disclosed, it may be required to be redacted. Upon request by the study funder, the PI may be asked to withhold disclosure for an additional 90 days to allow the study funder to seek patent protection.